CLINICAL TRIAL: NCT06325839
Title: Effects of HypnoBirthing Training and Oxytocin Massage on Delivery and Postpartum Period in Primiparous Pregnants: A Randomized Controlled Study
Brief Title: Effects of HypnoBirthing Training and Oxytocin Massage in Primiparous Pregnants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, ezgi.sahin, Assıstant Professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GRU-SBF-ES-01
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Birth; oxytocin; postpartum; hypno-birthing

STUDY DESIGN:
Intervention Model Description: The research is an experimental study with a randomized control group.
Who Masked: Participant
Masking Description: Pregnant women included in the study were randomly divided into two groups using the sealed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HypnoBirthing training and oxytocin massage group (Experimental): Pregnant women who received HypnoBirthing training and oxytocin massage constituted the experimental group.
  Interventions: Other: HypnoBirthing training and oxytocin massage group
- The group without HypnoBirthing training and oxytocin massage (No Intervention): Pregnant women who did not receive HypnoBirthing training and oxytocin massage constituted the control group.

INTERVENTIONS:
Other: HypnoBirthing training and oxytocin massage group — HypnoBirthing training and oxytocin massage were applied for a total of 12 hours for 4 weeks with the experimental group.
  Arms: HypnoBirthing training and oxytocin massage group

SUMMARY:
This study was conducted to determine the effects of hypnobirthing training and oxytocin massage on birth and postpartum period in primiparous pregnant women.

DETAILED DESCRIPTION:
Hypnobirthing is a birth philosophy and method that prepares women physically and psychologically for giving birth. It is important to break the fear-tension-pain cycle in HypnoBirthing training. Because the continuity of the cycle increases the pain related to birth, and as the pain increases, the fear increases. In this case, the duration of labor is prolonged, birth success, shape, preference, course and satisfaction are negatively affected. Therefore, this training helps to reduce pain and fear related to labor and increase labor satisfaction. Similarly, it has been determined in the literature that oxytocin (back massage) massage during pregnancy increases uterine contractions, reduces labor pain and duration of labor, accelerates postpartum uterine involution, significantly increases the amount of breast milk, and increases mother-baby attachment. The pregnant education role of the health professional is an effective factor that shapes the birth experience of pregnant women. For this purpose, health professionals in the world and in our country are actively involved in pregnancy education programs in which different methods are applied. The most common ones are Lamaze, Bradly and HypnoBirthing. These trainings also serve to reduce pain and fear related to childbirth, increase labor and postpartum satisfaction, and meet the need for professional support and education of pregnant women. When the studies on HypnoBirthing training and oxytocin massage are examined in the literature, it is noteworthy that there is a very limited number of studies. Therefore, there is a need for well-designed randomized controlled trials that can create a level of evidence for HypnoBirthing training and oxytocin massage.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18 and 45,
* Able to communicate verbally,
* Being in the 36th week of pregnancy,
* Having a single fetus,
* Being nulliparous

Exclusion Criteria:

* Pregnant women at risk
* Multiparous pregnant women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Wijma Birth Anticipation/Experience Scale A (W-DEQ-A) | five weeks
  The WDEQ A is a six-point Likert-type scale consisting of 33 items, scored 0-5, with 0 being "completely" and 5 being "not at all". The pregnant woman is asked to indicate a number between 0 and 5 that suits her. W-DEQ-A scores were categorized into four subgroups. These are women with a low degree of fear of childbirth (W-DEQ-A score ≤37), women with moderate fear of childbirth (W-DEQ-A score between 38-65), women with severe fear of childbirth (W-DEQ-A score 66-84) and women with clinical fear of childbirth (W-DEQ-A score ≥ 85).

SECONDARY OUTCOMES:
Wijma Birth Expectancy/Expectation Scale B (W-DEQ-B) | Five weeks
  The scale consists of 33 items. The responses in the scale are numbered from 0 to 5 and are in six-point Likert type. 0 means "completely" and 5 means "not at all". The minimum score on the scale is 0, while the maximum score is 160. As the score increases, the fear of childbirth experienced by women increases.
Postpartum Breastfeeding Self-Efficacy Scale - Short Form | 5 weeks
  The scale consists of 14 items. The scale is a 5-point Likert scale, ranging from never sure (1 point) to always sure (5 points). The minimum score is 14 and the maximum score is 70. The scale has no cut-off point and a higher score means higher breastfeeding self-efficacy.
Mother-Infant Attachment Scale (MICS) | 5 weeks
  This scale, consisting of 8 items, is designed to be applied from the first day after birth and allows the mother to express her feelings towards her baby with a single word. It is a 4-point Likert scale. Responses consisting of four options are scored between 0-3, the lowest score that can be obtained from the scale is 0 and the highest score is 24. High scores indicate that mother-baby attachment is strong.
Birth satisfaction scale short form (BSS-SF) | 5 weeks
  BSS-SF is a 10-item scale of 5-point Likert type. The lowest score from the scale is "0" and the highest score is "40", and as the score obtained from the scale increases, the level of satisfaction increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi ŞAHİN, ph.D, Principal Investigator — Giresun University Faculty of Health Sciences
Locations (1):
- Giresun Gynecology and Children's Diseases Hospital, Giresun, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No